CLINICAL TRIAL: NCT01719887
Title: Effectiveness and Cost-effectiveness of Surgical Treatment of Humeral Shaft Fractures. Randomized Controlled Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Töölö Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Lasse Rämö, MD, PhD, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS-118/13/03/02/2012
Record Dates: First submitted 2012-10-28; First posted 2012-11-01 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Fracture
Keywords: humerus; humeral; shaft; diaphysis; fracture; RCT
MeSH Terms: conditions — Fractures, Bone | interventions — Conservative Treatment; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative treatment (Active Comparator): Conservative treatment with functional brace and physiotherapy.
  Interventions: Device: Conservative treatment; Other: Physiotherapy
- Operative treatment (Experimental): Operative treatment with open reduction and internal fixation with 4,5mm locking compression plate. Physiotherapy at 3 and 9 wks.
  Interventions: Procedure: Operative treatment; Other: Physiotherapy

INTERVENTIONS:
Device: Conservative treatment — Conservative treatment with functional brace.
  Arms: Conservative treatment
Procedure: Operative treatment — Operative treatment with open reduction and internal fixation using 4,5mm locking compression plate.
  Arms: Operative treatment
Other: Physiotherapy — Physiotherapy is arranged to both groups at 3 and 9 wks.

SUMMARY:
Humeral shaft fractures represent 1-3% of all fractures and 20% of the humeral fractures. These fractures have historically been treated mainly conservatively with good results. Recent development in fracture treatment and findings that certain fracture types are more prone to non-union and bracing-related functional problems of adjacent joints are somewhat common have caused increasing interest in treating these fractures surgically. Return to activities is also considered to be quicker among surgically treated patients.

The purpose of this study is to evaluate effectiveness and cost-effectiveness of surgical treatment of humeral shaft fractures. Patients with an unilateral humeral shaft fracture who are willing to participate in the study after informed consent are randomly assigned to two different treatment methods:

1. Surgical treatment with an open reduction and internal fixation with a 4,5mm locking plate.
2. Conservative treatment with functional bracing

The randomization is done using blocked randomization (block sizes are not known by the enrolling or assigning physician) and stratification is done according to fracture type (AO-OTA type A vs. type B/C) and radial nerve status (total/subtotal motor palsy vs. no palsy).

Standard follow-up visits at 6 weeks, 3, 6 and 12 months are arranged. Later follow-up visits are arranged at 2, 5 and 10 years for the study purpose. Patients fill evaluation forms and clinical and radiological assessments are made. The physiotherapist doing objective functional measurements is blinded to treatment method. Both study groups receive physiotherapy after the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old patient who agrees to the consent to participation in this study
* Unilateral dislocated humeral shaft fracture (dislocation over thickness of the bone cortex, fracture below the level of insertion of pectoralis major muscle and 5 cm above the olecranon fossa)
* Randomization can be done within 10 days and operation within 14 days after the initial trauma
* Patient is willing to participate all follow-up visits

Exclusion Criteria:

* Bilateral humeral shaft fracture
* A significant concomitant trauma of the same upper extremity that warrants operative treatment (fracture, tendon injury, soft tissue trauma)
* Other fracture or abdominal/thoracal trauma that warrants operative treatment
* Open fracture
* Pathological fracture
* Multi-trauma patient
* Vascular injury
* Plexus injury
* Previous trauma in the same upper extremity that causes functional deficit
* Trauma or condition that warrants use of walking aid (crutches, wheelchair etc)
* Disease that affects significantly general condition of the patient
* Significantly impaired ability to co-operate for any reason (substance abuse, mental disorder, dementia)
* Unwilling to accept both treatment methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-11-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand Score (DASH) | at 12 months

SECONDARY OUTCOMES:
Subjective assessment of the function of the upper extremity | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
  Numerical Rating Scale (NRS) 0-10
Constant Score | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
Elbow ROM | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
Health-related quality of life (15D) | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
Complications | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
  Incidence of complications (i.e. non-union, malunion, re-fracture, reoperation, infection and iatrogenic radial palsy) is recorded and compared between study groups.
Cost-effectiveness | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
  Quality-adjusted life years/months measured as a change in 15D tool, pain-NRS and other outcome measures.
Subjective assessment of the function of the upper extremity | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
  Likert Scale 1-7
Subjective assessment of the function of the elbow | 6 wks, 3, 6, 12 mo, 2, 5, 10 years
  Numerical Rating Scale (NRS) 0-10
The Disabilities of the Arm, Shoulder and Hand Score (DASH) | at 6 wks, 3, 6 mo, 2, 5, 10 years
Pain at rest and in activity, Numerical Rating Scale (NRS) 0-10 | at 6 wks, 3, 6 mo, 12 mo, 2, 5, 10 years
Percentage of patients with acceptable symptom state (PASS) | at 6 wks, 3, 6 mo, 12 mo, 2, 5, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mika Paavola, MD, PhD, Study Director — Töölö Hospital
Locations (2):
- Finland (2):
  - Töölö Hospital, Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere

REFERENCES:
- [Background] Ramo L, Taimela S, Lepola V, Malmivaara A, Lahdeoja T, Paavola M. Open reduction and internal fixation of humeral shaft fractures versus conservative treatment with a functional brace: a study protocol of a randomised controlled trial embedded in a cohort. BMJ Open. 2017 Jul 9;7(7):e014076. doi: 10.1136/bmjopen-2016-014076. PMID 28694341
- [Result] Ramo L, Sumrein BO, Lepola V, Lahdeoja T, Ranstam J, Paavola M, Jarvinen T, Taimela S; FISH Investigators. Effect of Surgery vs Functional Bracing on Functional Outcome Among Patients With Closed Displaced Humeral Shaft Fractures: The FISH Randomized Clinical Trial. JAMA. 2020 May 12;323(18):1792-1801. doi: 10.1001/jama.2020.3182. PMID 32396179
- [Result] Ramo L, Paavola M, Sumrein BO, Lepola V, Lahdeoja T, Ranstam J, Jarvinen TLN, Taimela S; FISH Investigators. Outcomes With Surgery vs Functional Bracing for Patients With Closed, Displaced Humeral Shaft Fractures and the Need for Secondary Surgery: A Prespecified Secondary Analysis of the FISH Randomized Clinical Trial. JAMA Surg. 2021 Apr 14;156(6):1-9. doi: 10.1001/jamasurg.2021.0906. Online ahead of print. PMID 33851991
- [Result] Ramo L, Ibounig T, Sumrein BO, Lepola V, Paavola M, Taimela S, Jarvinen TLN; FISH Investigators. Five-Year Follow-Up of Surgery vs Functional Bracing for Closed Displaced Humeral Shaft Fractures. JAMA. 2024 Apr 2;331(13):1149-1151. doi: 10.1001/jama.2024.2671. PMID 38436996
- [Derived] Ibounig T, Juurakko J, Lahdeoja T, Sumrein BO, Jarvinen TLN, Paavola M, Ardern CL, Karjalainen T, Taimela S, Ramo L. Minimal important difference and patient acceptable symptom state for common outcome instruments in patients with a closed humeral shaft fracture - analysis of the FISH randomised clinical trial data. BMC Med Res Methodol. 2022 Nov 10;22(1):291. doi: 10.1186/s12874-022-01776-6. PMID 36357855